CLINICAL TRIAL: NCT02765191
Title: MR-Evaluation of Renal Function In Septic Patients
Acronym: MERSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MERSEP-523-2014-2569
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Sepsis, Severe; Acute Kidney Injury; COVID-19
Keywords: Magnetic Resonance Imaging; Fluid Therapy; Renal Circulation; Renal Oxygenation
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; COVID-19 | interventions — Ringer's acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Subjects investigated according to protocol after administration of bolus of Ringer's Acetate
  Interventions: Other: Plasma expansion with Ringer's Acetate

INTERVENTIONS:
Other: Plasma expansion with Ringer's Acetate — 7,5 ml/kg mL Ringer's acetate during 5-10 minutes will be administered intravenously

SUMMARY:
A study of renal blood flow and renal oxygenation measured by magnetic resonance after a standardized fluid challenge in critically ill, resuscitated, patients with sepsis due to COVID-19 or other agents.

DETAILED DESCRIPTION:
Critically ill, septic patients with or without acute kidney injury (AKI) above 18 years of age who have been circulatory and respiratory stabilized will be screened for inclusion.

After the patients have been adequately treated with antimicrobial agents, source control and circulatory and respiratory stabilized, the patient will be moved to the Magnetic resonance imaging (MRI)-suite and placed in the MRI-camera. We plan to, at the same time, study renal blood flow (RBF) and oxygenation with 4 different MRI techniques; arterial spin labeling (ASL), Blood oxygen level dependent (BOLD)-technique, T(2) -Relaxation-Under-Spin-Tagging (TRUST) and Phase contrast at two conditions;

1. at baseline after stabilization
2. after intravenous infusion of 7,5 ml/kg mL Ringer's acetate

The following data will be registered:

1. Age, gender, length and weight,
2. concomitant diseases and treatment,
3. present disease and treatment,
4. source of admission - emergency department or ordinary ward,
5. daily laboratory reports,
6. results from other investigations, e.g. x-rays, cultures etc.,
7. recordings from the intensive care unit (ICU) monitors
8. Continuous renal replacement therapy (CRRT) - duration type, flow rate, replacement fluid, etc.
9. dead or alive at discharge and 90 days mortality,
10. renal function at discharge,
11. treatment restrictions,
12. if the patient has died, the results from a possible postmortem examination. As well as all data obtained during the MRI-examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis sepsis (infection and organ dysfuncion) treated in intensive care.
* Manifest Acute kidney injury (AKI) or risk of AKI.
* 18 years of age or older

Exclusion Criteria:

* Pregnancy
* Chronic kidney failure
* Renal Replacement Therapy
* Instability in vital parameters to a degree where MRI is not feasible
* Contraindications for MRI (implants, coils, pacemakers, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Change in renal blood flow and renal oxygenation after standardized plasma expansion with fluid bolus | When achieved according to protocol, approximately 3-10 minutes after intervention
  Measured with arterial spin labelling (ASL), Phase Contras, Blood oxygenation level dependent (BOLD) and T(2) -Relaxation-Under-Spin-Tagging (TRUST), compared to baseline measurement
Descriptive renal oxygenation and blood flow in critical illness due to sepsis | During Critical illness - at one time point
  Measured with arterial spin labelling (ASL), Phase Contras, Blood oxygenation level dependent (BOLD) and T(2) -Relaxation-Under-Spin-Tagging (TRUST) during baseline measurement.
Descriptive renal oxygenation and blood flow in critical illness in no/low grade AKI or high grade AKI. | During Critical illness - at one time point
  Measured with arterial spin labelling (ASL), Phase Contras, Blood oxygenation level dependent (BOLD) and T(2) -Relaxation-Under-Spin-Tagging (TRUST) images stratified in groups in regards to KDIGO grade during exam.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frithiof, Assoc. Prof., Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luther T, Eckerbom P, Cox E, Lipcsey M, Bulow S, Hultstrom M, Torrente FM, Weis J, Palm F, Francis S, Frithiof R, Liss P. Decreased renal perfusion during acute kidney injury in critical COVID-19 assessed by magnetic resonance imaging: a prospective case control study. Crit Care. 2022 Sep 1;26(1):262. doi: 10.1186/s13054-022-04132-8. PMID 36050748